CLINICAL TRIAL: NCT07058415
Title: Osteoarticular Infections on Equipment: Impact of Three Probabilistic Antibiotic Therapy on Digestive Microbiota and Colonization With Multi-resistant Bacteria
Brief Title: Impact of Three Probabilistic Antibiotic Therapy on Digestive Microbiota and Colonization With Multi-resistant Bacteria
Acronym: HOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-CONS-01
Record Dates: First submitted 2025-03-10; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Osteoarticular Material Infection

STUDY DESIGN:
Intervention Model Description: Comparative, randomized, multicentric clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Céfépime + Daptomycine (Active Comparator): First stool sample taken the day before starting antibiotic therapy. Second stool sample on the fourth post-operative day (D5). Third stool sample taken 28 days after the end of antibiotic treatment (DX+28).
  Interventions: Other: Stool sample 1; Other: Stool sample 2; Other: Stool sample 3
- Pipéracilline-Tazobactam + Daptomycine (Active Comparator): First stool sample taken the day before starting antibiotic therapy. Second stool sample on the fourth post-operative day (D5). Third stool sample taken 28 days after the end of antibiotic treatment (DX+28).
  Interventions: Other: Stool sample 1; Other: Stool sample 2; Other: Stool sample 3
- Ceftobiprole (Experimental): First stool sample taken the day before starting antibiotic therapy. Second stool sample on the fourth post-operative day (D5). Third stool sample taken 28 days after the end of antibiotic treatment (DX+28).
  Interventions: Other: Stool sample 1; Other: Stool sample 2; Other: Stool sample 3

INTERVENTIONS:
Other: Stool sample 1 — Stool sampling at D0 for having baseline reference
Other: Stool sample 2 — Stool sampling at D5 to study the impact of antibiotics on microbiota
Other: Stool sample 3 — Stool sampling at DX+28 to study the impact of antibiotics on microbiota

SUMMARY:
In the event of suspected osteoarticular material infection (OAMI), broad-spectrum probabilistic antibiotic therapy is recommended immediately after revision surgery. There are no efficacy data to suggest that any particular to favour any particular molecule. However, the choice may depend on the impact on the microbiota and on Enterobacteriaceae colonization with multi-resistant Enterobacteriaceae. Our aim is to evaluate three different strategies efepime+daptomycin C+D, piperacillin-tazobactam+daptomycin (PT+D) and ceftobiprole (CFB).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for prosthetic revision (PTG, PUC, PTH or hip hemiarthroplasty, PTE) or internal osteosynthesis with suspicion of IOAM following the opinion of a Réunion de concertation Pluridisciplinaire (RCP) on complex osteoarticular infections
* Normal CPK level according to laboratory standard
* Social security affiliation
* Signature of informed consent
* Negative pregnancy test for women of childbearing age.

Exclusion Criteria:

* Antibiotic therapy in the 3 months prior to inclusion
* Clinical or radiological signs making HAI highly probable: scar discharge and/or peri-scar cellulitis fistula or abscess, bacteremia
* positive bacterial culture from joint puncture or biopsy prior to revision
* Chronic inflammatory bowel disease.
* Previous surgical resection of small intestine or colon.
* Hypersensitivity to daptomycin or any of its excipients.
* Hypersensitivity to cefepime or any of its excipients or to other beta-lactamins.
* Hypersensitivity to piperacillin+tazobactam or to any of the excipients or to other beta-lactamines.
* Hypersensitivity to ceftobiprole or to any of the excipients or to other beta-lactamines.
* Renal insufficiency with GFR < 50ml/min/1.73 m2 (CKD-EPI).
* Treatment with bosentan.
* Treatment with probenecid.
* Pre-existing seizure disorder.
* Contraindication to L-arginine, acidosis, hyperkalemia that cannot be corrected.
* Treatment with HMG-CoA reductase inhibitors.
* Treatment with statins (pitavastin, pravastatin, rosuvastatin) or glyburide.
* Patients in a medical emergency.
* Pregnant or breast-feeding women.
* Patient participating in another ongoing trial.
* Mental state rendering the patient incapable of understanding this research.
* Patient deprived of liberty by administrative or judicial decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Compare changes in gut microbiota biodiversity between Day1 and Day5 between populations treated with C+D, PT+D and CFB in suspected Osteoarticular infection on equipment | At Day 5 after starting treatment
  using targeted metagenomics (16S rDNA)

SECONDARY OUTCOMES:
Compare the evolution between Day1/end of treatment+28 Days and between Day 5/end of treatment+28D of microbiota biodiversity of each patient population treated with different antibiotics for suspected Osteoarticular infection on equipment | Up to 4 months
  Simpson index,
Compare the rate of acquisition of multidrug-resistant extended-spectrum beta-lactamase-producing intestinal Enterobacteria between antibiotic strategies on samples at Day5 and DX+28 in patients with no multidrug-resistant Enterobacteria at Day1. | Up to 4 months
  Stool culture on a selective medium at Day1, Day5 and Day X+28
Compare the rate of acquisition of carbapenemase-producing intestinal multi-resistant Enterobacteriaceae (EPC) between antibiotic strategies on samples taken at D5 and DX+28 in patients with no multi-resistant Enterobacteria at D1. | Up to 4 months
  The appearance of EPC-type multi-resistant Enterobacteriaceae will be determined by stool culture on a selective medium selective medium (mSuperCARBA, MAST diagnostic) at D1, D5 and DX+28.
Comparison of the rate of inadequacy of probabilistic strategies in the event of retained infection. | Up to 4 months
  Inadequacy of one of the three probabilistic strategies will be defined by a documented infection with a bacterium resistant to both antibiotics in the case of dual therapy, or to ceftobiprole in the case of monotherapy.
Compare the evolution between J5/JX+28 of microbiota biodiversity of patients receiving no antibiotic treatment for infection and patients in whom an infection is detected, with antibiotic treatment prescribed for 6 to 12 weeks. | Up to 4 months
  Shannon index
Compare the evolution between J5/JX+28 of microbiota biodiversity of patients receiving no antibiotic treatment for infection and patients in whom an infection is detected, with antibiotic treatment prescribed for 6 to 12 weeks. | Up to 4 months
  Piélou equitability index

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Ch Antibes, Antibes
  - Ch Cannes, Cannes
  - Ch Grasse, Grasse
  - CHU de NICE, Nice

IPD SHARING:
Plan to Share IPD: No